CLINICAL TRIAL: NCT06574503
Title: A Phase III, Multicenter, Randomized, Double-blind, Placebo-controlled, Clinical Efficacy and Safety Study of GP681 Tablets for Post-exposure Prophylaxis Against Influenza in Adults and Adolescents
Brief Title: Study to Assess the Efficacy and Safety of GP681 Versus Placebo for Postexposure Prophylaxis Against Influenza
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangxi Qingfeng Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GP681-202403
Record Dates: First submitted 2024-08-25; First posted 2024-08-28 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GP681 tablet 40mg (Experimental): atients in the GP681 tablet 40mg group will receive a single oral dose of GP681 tablet 40mg with water.
  Interventions: Drug: GP681 40mg
- Placebo group (Placebo Comparator): Patients in the Placebo group will receive a single oral dose of GP681 Simulant 40mg with water.
  Interventions: Drug: GP681 Simulant

INTERVENTIONS:
Drug: GP681 40mg — 2X20mg tablets taken orally
  Arms: GP681 tablet 40mg
Drug: GP681 Simulant — Placebo tablets matching GP681 40mg
  Arms: Placebo group

SUMMARY:
Index patients who are infected with influenza virus (Q-PCR positive) can be treated with anti-influenza drugs if their influenza symptoms onset was within 48 hours of screening. Their eligible households will be randomized to either GP681 tablets or placebo if at least 1 household contacts have not received influenza vaccine with 6 months of screening and if all household contacts screen negative for influenza infection. The main endpoints are assessed based on multiple respiratory swabs, obtained from household contacts up to Day 10, and through the assessment of symptoms.

ELIGIBILITY:
Inclusion Criteria:

Index patients(IPs)

1. Male or female patients aged≥2 years at the time of signing the informed consent form.
2. The first patient in a household with a diagnosis of influenza virus infection confirmed by all of the following in the influenza season:
3. Positive Influenza rapid antigen test or Polymerase chain reaction (PCR), and;
4. Fever (axillary temperature ≥37.3℃) in the predose examinations or > 4 hours after dosing of antipyretics if they were taken.
5. Patients with onset of fever within 48 hours or less at informed consent.
6. Patients live in a household where all household contacts are expected to meet the key household contacts inclusion criteria (criteria 2, 3, & 4).
7. Patients and/or their guardian who are willing to provide written informed consent and consent to participate in the study, able to understand the study and comply with all study procedures.

Household contacts of index patients:

1. Male or female patients aged≥12 years at the time of signing the informed consent form.
2. Household contacts who are able to provide informed consent within 24 hours or less from informed consent in index patients.
3. Subjects who had lived with the index patient for 3 months or more prior to informed consent.
4. Subjects who meet all of the following criteria and are judged not to have influenza virus infection by the investigator.
5. Negative Influenza rapid antigen test or Polymerase chain reaction (PCR), and;
6. Subjects who have a body temperature (axillary) < 37.3°C at Screening, and;
7. Subjects who have no influenza like symptoms (cough, sore throat, headache, nasal discharge/nasal congestion, feverishness or chills, muscle or joint pain, and fatigue) at Screening.
8. Household contacts intended for full study have not received influenza vaccine within 6 months prior to screening;
9. Subjects and/or their guardian who are willing to provide written informed consent and consent to participate in the study, able to understand the study and comply with all study procedures, including patient health diary records.

Exclusion Criteria:

Household contacts of index patients:

1. History of allergic reactions attributed to GP681 or any of the ingredients of its formulation.
2. Subjects with household members other than the index patient that was diagnosed with or strongly suspected to have influenza in the past 12 weeks.
3. subjects with concurrent bacterial or other virus infections requiring systemic antimicrobial and/or antiviral therapy at the pre-dose examinations.
4. Subjects who are unable to live with the index patient from Screening until Day 10.
5. Known history of dysphagia or any gastrointestinal disease that affects drug absorption (including but not limited to reflux esophagitis, chronic diarrhea, inflammatory bowel disease, intestinal tuberculosis, gastrinoma, short bowel syndrome, stomach after subtotal resection, etc.).
6. Subjects who have any underlying diseases requiring systemic , treatment of antipyretics/analgesics, corticosteroids, or immunosuppressive agents.
7. Subjects with human immunodeficiency virus [HIV] infection.
8. Subjects with severe (Grade 3 or higher of Common Terminology Criteria for Adverse Events [CTCAE] ver. 5) underlying diseases.
9. Treatment with anti-influenza virus drugs (oseltamivir, zanamivir, peramivir, favipiravir, abidol, baloxavir marboxil, amantadine, or rimantadine) within 2 weeks before screening.
10. Known history of alcohol abuse (Average weekly intake of alcohol is more than 14 units alcohol (1 units ≈ 360 mL beer, or 45 mL spirits with 40% content, or 150 mL wine) or drug abuse at screening;
11. Women who are pregnant, breastfeeding, or have a positive pregnancy test at the predose examinations. The following female patients who have documentation of either a or below do not need to undergo a pregnancy test at the predose examinations:

    1. Postmenopausal women (defined as cessation of regular menstrual periods for 2 years or more and aged more than 50 years old)
    2. Women who are surgically sterile by hysterectomy, bilateral oophorectomy, or tubal ligation
12. Has received any investigational agents or devices for any indication within 30 days prior to Screening.
13. Subjects who, in the opinion of the Investigator, may not be qualified or suitable for the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 748 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of household members who are infected with influenza virus (Q-PCR positive), and present with fever and at least one influenza symptom with severity of moderate or severe in the period from Day 1 to Day 10. | up to Day 10
  Defined as the proportion of household members having body temperature (axillary)≥37.3°C, having symptom of influenza (respiratory symptoms or systemic symptoms) with a severity of "2, Moderate" or "3, Severe" assessed in the subject diary, and influenza virus positive assessed by Q-PCR.

SECONDARY OUTCOMES:
Proportion of household members who are infected with influenza virus (Q-PCR positive), and present with fever or at least one influenza symptom with severity of moderate or severe in the period from Day 1 to Day 10. | up to Day10
  Defined as the proportion of household members having body temperature (axillary)≥37.3°C, or having symptom of influenza (respiratory symptoms or systemic symptoms) with a severity of "2, Moderate" or "3, Severe" assessed in the subject diary, and influenza virus positive assessed by Q-PCR.
Proportion of household members with influenza virus infection in the period from Day 1 to Day 10 | up to Day10
  Defined as the proportion of subjects having influenza virus positive assessed by RT-PCR regardless of body temperature or influenza symptoms.
Time from study treatment to the time when fever, at least one influenza symptom with severity of moderate or severe, and influenza virus infection were observed. | up to Day10
  Defined as the later timepoint of the following (1) and (2):
  1. Timepoint when body temperature (axillary) rises first to " 37.3°C
  2. Timepoint when an influenza symptom was first assessed as"2, Moderate" or "3, Severe" in the subject diary.
  If a household member does not have a body temperature (axillary) of "37.3°C or influenza symptom was not assessed as"2, Moderate" or "3, Severe" in the period from Day 1 to Day 10, the subject will be handled as a censored case.
Time from study treatment to the time when fever or at least one influenza symptom (respiratory symptom or systemic symptom), and influenza virus infection are observed. | up to Day10
  Defined as the timepoint of the following (1) and (2), whichever is earlier:
  1. Timepoint when body temperature (axillary) rises first to " 37.3°C
  2. Timepoint when an influenza symptom was first assessed as"2, Moderate" or "3, Severe" in the subject diary.
  If a subject does not have a body temperature (axillary) of "37.5°C and influenza symptoms (respiratory symptoms and systemic symptoms) were not assessed as 2, Moderate or 3, Severe in the period from Day 1 to Day 10, the subject will be handled as a censored case.
Proportion of asymptomatic influenza-infected (Q-PCR positive) household members in the period from Day 1 to Day 10 | Up to Day 10
  Defined as the proportion of household members having body temperature (axillary) < 37.5°C, influenza symptoms all assessed as 0, Absent or 1, Mild , and influenza virus positive assessed by Q-PCR.
Proportion of household members who are not infected with influenza virus (Q-PCR negative) and present with fever and at least one influenza symptom with severity of moderate or severe in the period from Day 1 to Day 10 | Up to Day 10
  Defined as the proportion of household members having body temperature (axillary) "37.3°C, having symptom of influenza (respiratory symptoms or systemic symptoms) with a severity of "2, Moderate" or "3, Severe" assessed in the subject diary, and influenza virus negative at all time points assessed by Q-PCR.
Proportion of household members who are infected with influenza virus (Q-PCR positive) in the period from Day 1 to Day 10, with virus subtype consistent with index patient | Up to Day 10
  Defined as the proportion of household members who are infected with influenza virus (Q-PCR positive) in the period from Day 1 to Day 10，and the virus subtype of household members are consistent with index patient

CONTACTS AND LOCATIONS:
Locations (1):
- Shulan (Hang Zhou) Hospital, Hanzhou, China

IPD SHARING:
Plan to Share IPD: No